CLINICAL TRIAL: NCT05045885
Title: Safety and Feasibility of Percutaneous Dilatational Tracheostomy in Patients With Severe COVID-19 Disease Supported by Extracorporeal Membrane Oxygenation.
Brief Title: Safety and Feasibility of Percutaneous Dilatational Tracheostomy in Patients With Severe COVID-19 Supported by ECMO
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-20-1196
Record Dates: First submitted 2021-09-14; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Pneumonia; Extracorporeal Membrane Oxygenation Complication; Tracheostomy Complication; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 pandemic has presented the global health care systems with unprecedented and unexpected challenges. The clinical spectrum of COVID-19 disease varies from mild, at times asymptomatic, to severe life-threatening multiple organ dysfunction and shock. The latter group, albeit represent less than 10% of all SARS-CoV-2 infections will require ICU admission, multi-modal organ support including Extracorporeal Membrane Oxygenation (ECMO) for severe refractory cardiac and/or pulmonary failure.

Prolonged mechanical ventilation is a typical indication for tracheostomy. Percutaneous tracheostomy at the bedside has several advantages over surgical tracheostomy. However, with the emerging pandemic, there is a lack of literature regarding the safety of percutaneous bedside tracheostomy for patients with COVID-19 supported by ECMO.

Our study aims to describe the safety of bedside percutaneous dilatational tracheostomy of confirmed COVID-19 positive patients supported on ECMO.

DETAILED DESCRIPTION:
At the time of writing, more than 50 million confirmed cases of COVID-19 have been reported worldwide with over one million reported deaths1 Data about ICU mortality is variable and may be affected by the infrastructure of the health care system in each country, however, the estimated mortality rate in COVID-19 patients who need ICU is 25.7%-35.7%2.

The World Health Organization (WHO) suggests ECMO for COVID-19 patients with severe ARDS not responding to conventional treatment. However, Extracorporeal Life Support Organization (ESLSO) guidance recommends a balance of resource utilization, allocation, and appropriate case selection3.

According to ELSO Registry; 3048 COVID-19 cases have been supported on ECMO. Interestingly discharge alive rate was reported to be over 60%4.

Tracheostomy can be performed with two different techniques. Open 'surgical' tracheostomy (OT) and percutaneous dilatational tracheostomy (PDT). The later was favored during the SARS outbreak (SARS-CoV-1). However, the literature is not clear yet about the preferable and safest technique during Covid-19 disease SARS-CoV-2 as both procedures could be aerosol-generating procedures (AGP)5,6.

SARS-CoV-2 is highly contagious and can spread via aerosol, contact, and droplet. This poses a significant risk to health care workers (HCW) and in particular during airway interventions and procedures.

The optimal time to perform tracheostomy in COVID-19 patients remains controversial. Recommendations are different whether early or late tracheostomy is the preferred one, however, the American Academy of Otolaryngology-Head and Neck surgery recommend the procedure to take a place 2-3 weeks after intubation5,6.

Generally speaking, tracheostomy has many advantages in critically ill patients such as reducing the days of mechanical ventilation, reduce ICU admission, reduce nosocomial pneumonia in special groups7,8.

Tracheostomy carries the second-highest risk of transmission of infection to staff after endotracheal intubation. PDT in patients supported on ECMO is not without risks. Bleeding is a major concern and has been reported at 40%9-11. Other reported procedural complications are mechanical and ECMO-circuit dysfunction9-12.

The literature search revealed one case series from the UK13 of PDT in the same patient population as our study. However, the report focuses on the description of the procedure rather than the safety aspect. To my knowledge, this is the first study to look in-depth into staff and patient safety of PDT in COVID-19 positive patients on ECMO support.

ELIGIBILITY:
Inclusion Criteria:

* over 18-years old.

Exclusion Criteria:

* less than 18 years old,
* Pregnancy
* VA-ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The COVID and non-COVID patients on VV ECMO who underwent percutaneous dilatational tracheostomy (PDT).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
External or endotracheal bleeding (mild, moderate, sever) | 24 hours Post procedure
  Mild: Minimal external or endotracheal bleeding with minimal or no drop-in haemoglobin and no surgical intervention.
  Moderate: Obvious external or endotracheal bleed. A drop-in haemoglobin of less than one gram/dL or transfusion of one unit of red blood cells.
  Severe bleeding: a drop of two grams or more in haemoglobin/dL and/or transfusion of two or more red cell packs or other blood products, disseminated intravascular coagulopathy (DIC) or need for surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Labib, Principal Investigator — Hamad Medical Corporation - HMC
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
After approval of Hospital IRB
Supporting Information: Study Protocol
Time Frame: After finishing the study
Access Criteria: Website

REFERENCES:
- [Background] WHO Director-General's opening remarks at the media briefing on COVID-19: 11 March 2020. Published March 11, 2020
- [Background] COVID Live Update: 189,294,523 Cases and 4,076,726 Deaths from the Coronavirus - Worldometer. Worldometers.info. https://www.worldometers.info/coronavirus/. Published 2021. Accessed July 15, 2021.
- [Background] Extracorporeal Life Support Organization - ECMO and ECLS. Elso.org. https://www.elso.org/COVID19.aspx. Published 2021. Accessed June 9, 2021.
- [Background] Tracheotomy Recommendations During the COVID-19 Pandemic - American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS). American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS). https://www.entnet.org/resource/tracheotomy-recommendations-during-the-covid-19-pandemic-2/. Published 2021. Accessed June 9, 2021.
- [Result] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Auld SC, Caridi-Scheible M, Blum JM, Robichaux C, Kraft C, Jacob JT, Jabaley CS, Carpenter D, Kaplow R, Hernandez-Romieu AC, Adelman MW, Martin GS, Coopersmith CM, Murphy DJ; and the Emory COVID-19 Quality and Clinical Research Collaborative. ICU and Ventilator Mortality Among Critically Ill Adults With Coronavirus Disease 2019. Crit Care Med. 2020 Sep;48(9):e799-e804. doi: 10.1097/CCM.0000000000004457. PMID 32452888
- [Result] Shekar K, Badulak J, Peek G, Boeken U, Dalton HJ, Arora L, Zakhary B, Ramanathan K, Starr J, Akkanti B, Antonini MV, Ogino MT, Raman L, Barret N, Brodie D, Combes A, Lorusso R, MacLaren G, Muller T, Paden M, Pellegrino V; ELSO Guideline Working Group. Extracorporeal Life Support Organization Coronavirus Disease 2019 Interim Guidelines: A Consensus Document from an International Group of Interdisciplinary Extracorporeal Membrane Oxygenation Providers. ASAIO J. 2020 Jul;66(7):707-721. doi: 10.1097/MAT.0000000000001193. PMID 32604322
- [Result] Nieszkowska A, Combes A, Luyt CE, Ksibi H, Trouillet JL, Gibert C, Chastre J. Impact of tracheotomy on sedative administration, sedation level, and comfort of mechanically ventilated intensive care unit patients. Crit Care Med. 2005 Nov;33(11):2527-33. doi: 10.1097/01.ccm.0000186898.58709.aa. PMID 16276177
- [Result] Dempsey GA, Grant CA, Jones TM. Percutaneous tracheostomy: a 6 yr prospective evaluation of the single tapered dilator technique. Br J Anaesth. 2010 Dec;105(6):782-8. doi: 10.1093/bja/aeq238. Epub 2010 Sep 2. PMID 20813838
- [Result] Beiderlinden M, Eikermann M, Lehmann N, Adamzik M, Peters J. Risk factors associated with bleeding during and after percutaneous dilational tracheostomy. Anaesthesia. 2007 Apr;62(4):342-6. doi: 10.1111/j.1365-2044.2007.04979.x. PMID 17381569
- [Result] Tang S, Mao Y, Jones RM, Tan Q, Ji JS, Li N, Shen J, Lv Y, Pan L, Ding P, Wang X, Wang Y, MacIntyre CR, Shi X. Aerosol transmission of SARS-CoV-2? Evidence, prevention and control. Environ Int. 2020 Nov;144:106039. doi: 10.1016/j.envint.2020.106039. Epub 2020 Aug 7. PMID 32822927
- [Result] Weissman DN, de Perio MA, Radonovich LJ Jr. COVID-19 and Risks Posed to Personnel During Endotracheal Intubation. JAMA. 2020 May 26;323(20):2027-2028. doi: 10.1001/jama.2020.6627. No abstract available. PMID 32338710
- [Result] Chorath K, Hoang A, Rajasekaran K, Moreira A. Association of Early vs Late Tracheostomy Placement With Pneumonia and Ventilator Days in Critically Ill Patients: A Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2021 May 1;147(5):450-459. doi: 10.1001/jamaoto.2021.0025. PMID 33704354
- [Result] Zangrillo A, Landoni G, Biondi-Zoccai G, Greco M, Greco T, Frati G, Patroniti N, Antonelli M, Pesenti A, Pappalardo F. A meta-analysis of complications and mortality of extracorporeal membrane oxygenation. Crit Care Resusc. 2013 Sep;15(3):172-8. PMID 23944202
- [Result] Braune S, Kienast S, Hadem J, Wiesner O, Wichmann D, Nierhaus A, Simon M, Welte T, Kluge S. Safety of percutaneous dilatational tracheostomy in patients on extracorporeal lung support. Intensive Care Med. 2013 Oct;39(10):1792-9. doi: 10.1007/s00134-013-3023-8. Epub 2013 Jul 27. PMID 23892417
- [Result] Kruit N, Valchanov K, Blaudszun G, Fowles JA, Vuylsteke A. Bleeding Complications Associated With Percutaneous Tracheostomy Insertion in Patients Supported With Venovenous Extracorporeal Membrane Oxygen Support: A 10-Year Institutional Experience. J Cardiothorac Vasc Anesth. 2018 Jun;32(3):1162-1166. doi: 10.1053/j.jvca.2017.08.010. Epub 2017 Aug 3. PMID 29129346
- [Result] Salna M, Tipograf Y, Liou P, Chicotka S, Biscotti M 3rd, Agerstrand C, Abrams D, Brodie D, Bacchetta M. Tracheostomy Is Safe During Extracorporeal Membrane Oxygenation Support. ASAIO J. 2020 Jun;66(6):652-656. doi: 10.1097/MAT.0000000000001059. PMID 31425269
- [Result] Dimopoulos S, Joyce H, Camporota L, Glover G, Ioannou N, Langrish CJ, Retter A, Meadows CIS, Barrett NA, Tricklebank S. Safety of Percutaneous Dilatational Tracheostomy During Veno-Venous Extracorporeal Membrane Oxygenation Support in Adults With Severe Respiratory Failure. Crit Care Med. 2019 Feb;47(2):e81-e88. doi: 10.1097/CCM.0000000000003515. PMID 30431492
- [Result] Valchanov K, Salaunkey K, Parmar J. Percutaneous Dilatational Tracheostomy in Coronavirus Disease 2019 Extracorporeal Membrane Oxygenation Patients: A Case Series. J Cardiothorac Vasc Anesth. 2021 Jan;35(1):348-350. doi: 10.1053/j.jvca.2020.06.024. Epub 2020 Jun 12. No abstract available. PMID 32620486
- [Result] Lamb CR, Desai NR, Angel L, Chaddha U, Sachdeva A, Sethi S, Bencheqroun H, Mehta H, Akulian J, Argento AC, Diaz-Mendoza J, Musani A, Murgu S. Use of Tracheostomy During the COVID-19 Pandemic: American College of Chest Physicians/American Association for Bronchology and Interventional Pulmonology/Association of Interventional Pulmonology Program Directors Expert Panel Report. Chest. 2020 Oct;158(4):1499-1514. doi: 10.1016/j.chest.2020.05.571. Epub 2020 Jun 6. PMID 32512006
- [Result] El Bouzidi K, Pirani T, Rosadas C, Ijaz S, Pearn M, Chaudhry S, Patel S, Sureda-Vives M, Fernandez N, Khan M, Cherepanov P, McClure MO, Tedder RS, Zuckerman M; COVID-STOICS (Serological Testing Of Intensive Care Staff). Severe Acute Respiratory Syndrome Coronavirus-2 Infections in Critical Care Staff: Beware the Risks Beyond the Bedside. Crit Care Med. 2021 Mar 1;49(3):428-436. doi: 10.1097/CCM.0000000000004878. PMID 33512941